CLINICAL TRIAL: NCT04377529
Title: Evaluating the Impact of a Champion on Implementation of the Back Skills Training (BeST) Program in Canada: a Mixed Methods Feasibility Study Protocol
Brief Title: Evaluating the Impact of a Champion on Implementation of the Back Skills Training (BeST) Program in Canada
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Amanda Hall, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20190025
Record Dates: First submitted 2020-04-22; First posted 2020-05-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
Keywords: implementation; behaviour change wheel; physiotherapy; cognitive behavioural therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Back Skills Training Champion (Experimental): In additional to access to the online provider Back Skills Training course, participants in clusters randomised to this arm will receive additional support from a local champion. The local champion will have received additional training and support on the implementation of the Back Skills Training intervention from the study team.
  Interventions: Behavioral: Local Champion
- No Champion (Active Comparator): Participants in clusters randomised to this arm will not receive any additional training or support beyond access to the online provider Back Skills Training course.
  Interventions: Behavioral: Local Champion

INTERVENTIONS:
Behavioral: Local Champion — Local champions (physiotherapists) will co-develop the champion training support based on a comprehensive behavioural analysis, previous implementation work and evidence-based theory. The study team will provide this training and support to the champions, who will then provide additional support to their peers participating in the study.

SUMMARY:
There is global recognition in clinical guidelines and governing bodies that low back pain (LBP) should be managed with a biopsychosocial approach. Despite this, research indicates that physiotherapists, who treat the majority of LBP patients in the community, do not feel confident in using this treatment approach. Previous work to support implementation in this field has resulted in low uptake and has highlighted several barriers to implementation, including the need for additional ongoing support. The use of a local champion to support implementation has been successful in other fields and thus, represents a viable strategy to explore. Before undertaking a fully powered trial to evaluate the effectiveness of a champion for implementation, a pilot study is being conducted to determine the feasibility of the intervention as well as determining the feasibility of using a cluster randomised controlled trial to evaluate it.

In this study, a pragmatic cluster randomised controlled trial design will be used with an embedded qualitative interview study. Physiotherapists will be recruited who manage LBP in any publicly funded physiotherapy departments within Newfoundland and Labrador, Canada. Individual sites will be grouped into clusters based on their number of full-time physiotherapists, geography, and organisational relationships. All participants will be asked to complete a previously developed online training course to upskill them to deliver a biopsychosocial evidence-based intervention for LBP. Clusters randomised to receive a local champion will receive additional support from their champion. A basic champion training package has been developed based on known barriers in the literature. This will be tailored by co-developing aspects with study champions based on a comprehensive assessment of perceived implementation barriers using the Theoretical Domains Framework (TDF) and the Capability, Opportunity, Motivation and Behaviour (COM-B) model. A range of physiotherapist-level outcomes pre-post training will be measured and implementation of the evidence based biopsychosocial intervention will be monitored during a 6-month period after completion of the online training. After this 6-month period, a purposive sample of physiotherapists from each cluster who had both implemented and failed to implement the biopsychosocial intervention will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Any publicly funded physiotherapy department within Newfoundland and Labrador working with adult patients with LBP are eligible to participate.
* Clinical leads need to be able to identify at least one champion at each site should they be allocated to the champion arm. We defined a champion as a physiotherapist in the musculoskeletal outpatient department who i) could commit the additional time for training, ii) would be willing to provide support to their peers at the sites within their cluster and iii) demonstrates enthusiasm about intervention to manager.

Exclusion Criteria:

* Physiotherapy departments who do not treat adult patients with LBP will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
% of target recruitment reached (champions) | 6 months post-intervention
  We aim to recruit at least 1 champion from each cluster.

SECONDARY OUTCOMES:
% of physiotherapists implementing the Back Skills Training intervention | 6-months post intervention
Qualitative analysis of barriers to both the champion training intervention and the Back Skills Training intervention | 6-months post intervention
  Individual semi-structured interviews
Satisfaction with champion training | Immediately post-intervention and at 6-months post-intervention
  A single item satisfaction score on a 5-point scale with 1=very unsatisfied and 5=very satisfied
Usefulness of the champion training | Immediately post-intervention and at 6-months post-intervention
  A single item usefulness score on a 5-point scale with 1=very unacceptable and 5=very acceptable
% of champions remaining at the end of the study follow-up period | 6-months post intervention
% of patients with low back pain who received the BeST intervention in each cluster | 6-months post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science Centre, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Derived] Hall A, Richmond H, Bursey K, Hansen Z, Williamson E, Copsey B, Albury C, Asghari S, Curran V, Pike A, Etchegary H, Lamb S. Evaluating the impact of a champion on implementation of the Back Skills Training (BeST) programme in Canada: a mixed methods feasibility study protocol. BMJ Open. 2020 Nov 30;10(11):e040834. doi: 10.1136/bmjopen-2020-040834. PMID 33257487